CLINICAL TRIAL: NCT06866405
Title: A Phase 3 Study to Investigate the Safety, Tolerability, and Immunogenicity of Revaccinating Pregnant Participants During Subsequent Pregnancies and Persistence of Immunity of a Single Dose of a Bivalent Respiratory Syncytial Virus (RSV) Vaccine.
Brief Title: A Phase 3 Study of Revaccination in Subsequent Pregnancies With Bivalent RSV Vaccine and Duration of Protection of a Single Dose
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671059; Marguerite (Other: Alias Study Number)
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: RSV Infection
Keywords: Pregnancy; RSV vaccine; RSV; Maternal immunization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding only applies to Cohort 2 of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RSVpreF (Experimental)
  Interventions: Biological: RSVpreF
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSVpreF — Single Dose
  Arms: RSVpreF
Biological: Placebo — Single Dose
  Arms: Placebo

SUMMARY:
This study aims to check how safe and well-tolerated a second dose of RSVpreF is when given during later pregnancies, and to see how long the immunity lasts from a single dose given during a previous pregnancy by examining the blood of nonpregnant participants who had the vaccine before.

DETAILED DESCRIPTION:
This study will include pregnant participants and their unborn babies (Cohort 1 and Cohort 2) and non-pregnant participants (Cohort 3), as described below:

* Cohort 1- Pregnant participants who had previously received RSVpreF as part of a Pfizer clinical trial and have antibody data available from that trial will get a second dose of RSVpreF.
* Cohort 2- Pregnant participants who received the RSVpreF in a previous pregnancy, either through commercial means with Abrysvo® or as part of a Pfizer clinical trial, will be randomly chosen to get either one dose of the RSVpreF or one dose of a placebo. This applies to those who do not have antibody data available from the earlier trial.

For both groups of pregnant participants, the study will look at how safe and well-tolerated the vaccine is during pregnancy, as well as how the body responds to it.

Infants will be monitored for six months after birth to check safety and antibodies level.

• Cohort 3- Nonpregnant participants who received RSVpreF during a previous pregnancy as part of an earlier clinical trial will have blood samples taken to see how well their immune response has persisted over time. Participants will not receive any vaccine.

ELIGIBILITY:
Pregnant Participants-Cohort 1 and Cohort 2 Key Inclusion Criteria

* Women aged 18 to 49 who are pregnant, between 24 and 36 weeks along, and expecting one baby without known risks for complications can participate.
* Had the RSVpreF or Abrysvo vaccine during a previous pregnancy.
* Had an ultrasound scan at 18 weeks or later during their current pregnancy, with no major fetal problems detected.
* Based on their medical history, physical check-up, and the doctor's judgment, they are found suitable to join the study.
* Agrees to let their baby take part in the study and gives their permission.
* Able to sign a consent form, agreeing to follow the rules and conditions of the study.

Key Exclusion Criteria

* Received any approved or experimental RSV vaccine since their previous pregnancy.
* Has a pre-pregnancy body mass index (BMI) over 40 kg/m2.
* History of a severe bad reaction to a vaccine or a serious allergic reaction (like anaphylaxis) to any ingredient in the study vaccine or a similar vaccine.
* Current pregnancy problems or issues at the time of giving consent.
* Previous pregnancy issues or problems at the time of giving consent.

Infant Participants

* Proof that the parent(s) or legal guardian(s) has signed and dated a consent form.
* Parent(s) or legal guardian(s) must agree to attend scheduled visits and follow the study plan, including laboratory tests and other procedures.

Nonpregnant Participants-Cohort 3 Key Inclusion Criteria

* Have already received one dose of the RSVpreF vaccine during their previous pregnancy as part of the Pfizer clinical trial, and the results from that time can be used for this study.
* Able to sign a consent form, agreeing to follow the rules and requirements of the study.

Key Exclusion Criteria

* Received any approved or experimental RSV vaccine after participating in the Pfizer clinical trial.
* Taking part in other studies with new drugs within 28 days before giving consent or during the study period.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2028-02-24 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of pregnant participants reporting local reactions | From Day 1 Through at least Day 7 after Vaccination
  Pain at the injection site, redness, and swelling
Percentage of pregnant participants reporting systemic events | From Day 1 Through at least Day 7 after Vaccination
  Fever, fatigue, headache, vomiting, nausea, diarrhea, muscle pain, and joint pain
Percentage of pregnant participants reporting adverse events | From Day 1 through 4 weeks after vaccination
Percentage of pregnant participants reporting serious adverse events | From Day 1 throughout the study
In infant participants born to pregnant participants receiving a second dose of the study intervention, the percentage of participants reporting adverse events. | From birth through 1 month of age
In infant participants born to pregnant participants receiving a second dose of the study intervention, the percentage of participants reporting serious adverse events and newly diagnosed medical conditions. | From birth through 6 months of age.
Proportion of participants achieving neutralizing antibody to RSV A and RSV B at birth | At birth

SECONDARY OUTCOMES:
Proportion of participants achieving neutralizing antibody to RSV A and RSV B at 3 months and 6 months | At 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (87):
- United States (75):
  - Center for Research in Women's Health, Birmingham, Alabama
  - Children's of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham - School of Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham Women & Infants Center, Birmingham, Alabama
  - USA Health Children's and Women's Hospital, Mobile, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Ronald Reagan UCLA Medical Center (inpatient hospital), Los Angeles, California
  - UCLA (outpatient clinic), Los Angeles, California
  - UCLA Clinical and Translational Research Center (research clinic), Los Angeles, California
  - UCLA, Los Angeles, California
  - Lucile Packard Children's Hospital-Labor and Delivery Unit, Palo Alto, California
  - Stanford Obstetrics Clinic, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - Stanford University, Palo Alto, California
  - Anschutz Health Sciences Building (AHSB), Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - CU Research Pharmacy, Aurora, Colorado
  - University of Colorado AO1 UCH, Aurora, Colorado
  - University of Colorado Hospital Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital Outpatient Pavilion, Aurora, Colorado
  - University of Colorado Research II Building, Aurora, Colorado
  - Citadelle Clinical Research, North Miami Beach, Florida
  - Emerald Coast OBGYN Clinical Research, Panama City, Florida
  - Emerald Coast Pediatrics, Panama City, Florida
  - HCA Florida Gulf Coast Hospital, Panama City, Florida
  - Emerald Coast Pediatrics, Panama City Beach, Florida
  - Advanced Specialty Research, Boise, Idaho
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Luke's Boise Medical Center, Boise, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Saint Alphonsus Medical Center, Nampa, Idaho
  - St. Luke's Nampa Medical Center, Nampa, Idaho
  - Accellacare - McFarland, Ames, Iowa
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic, PC, Ames, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - Velocity Clinical Research - New Orleans, New Orleans, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Velocity Clinical Research, Gulfport, Gulfport, Mississippi
  - Boeson Research GTF, Great Falls, Montana
  - OBGYN Associates, Great Falls, Montana
  - Boeson Research KAL, Kalispell, Montana
  - Heart & Hands Midwifery, Kalispell, Montana
  - Boeson Research MSO, Missoula, Montana
  - Origin Health, Missoula, Montana
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research, Norfolk, Norfolk, Nebraska
  - Presbyterian Hospital, Albuquerque, New Mexico
  - UNM Hospital, Albuquerque, New Mexico
  - Velocity Clinical Research, Albuquerque, Albuquerque, New Mexico
  - Lovelace Women's Hospital, Albuquerque, New Mexico
  - Duke University - Main Hospital and Clinics, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Prisma Health-Upstate, Greenville, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Memorial Hermann Memorial City Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Helios Clinical Research - WEA, Weatherford, Texas
  - Medical City Weatherford, Weatherford, Texas
  - Weatherford OB/GYN Associates, Weatherford, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Utah Clinical Neuroscience Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Sentara Leigh Hospital, Norfolk, Virginia
  - The Group For Women - Kempsville Office, Norfolk, Virginia
  - Tidewater Physicians for Women, Norfolk, Virginia
  - WomensCare Center, Norfolk, Virginia
  - Virginia Physicians For Women (VPFW), North Chesterfield, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Infusion Solutions, LLC, Richmond, Virginia
  - Seattle Children's Research Institute, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington - Northwest, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
- Argentina (7):
  - Fundación Respirar, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Clinica Del Niño Y La Madre, Mar del Plata, Buenos Aires
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Instituto de Maternidad y Ginecología Nuestra Señora de las Mercedes, San Miguel de Tucumán, Tucumán Province
  - Centro de investigación Clínica OSECAC - Sede Jonas Salk, Buenos Aires
  - Equipo Ciencia, Buenos Aires
  - Hospital Público Materno Infantil, Salta
- South Africa (5):
  - Josha Research, Bloemfontein, Free State
  - University of Witwatersrand (WITS) - Vaccines and Infectious Diseases Analytics (VIDA), Johannesburg, Gauteng
  - Wits RHI, Johannesburg, Gauteng
  - Into Research, Pretoria, Gauteng
  - MRC Unit on Child And Adolescent Health, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
Supporting Information: Study Protocol
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671059